CLINICAL TRIAL: NCT06780384
Title: NTRK 1,2,3 Rearrangements in Patients With Solid Tumors
Acronym: NTRK
Status: Active, not recruiting | Type: Observational
Sponsor: Federico Cappuzzo (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, Federico Cappuzzo, Professore Federico Cappuzzo, Fondazione Ricerca Traslazionale
Organization: Fondazione Ricerca Traslazionale (Other)
Other Study IDs: NTRK; NTRK (Other: Fondazionefort)
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: NTRK1/2/3 Fusion Gene Detection
Keywords: NTRK

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the incidence of NTRK rearrangements in patients with solid tumors in Italy. Additionally, the study seeks to define the correlation between IHC and FISH testing and to simplify the assessment of NTRK rearrangements in patients with solid tumors.

DETAILED DESCRIPTION:
Neurotrophic tropomyosin-related kinases (NTRKs, or the commonly used alias TRKs) constitute a receptor tyrosine kinase family of neurotrophin receptors involved in neuronal development, including the growth and function of neuronal synapses and memory development.

NTRK1/2/3 gene fusions have emerged as new targets for cancer therapy as they can be successfully inhibited by targeted kinase inhibitors. Several compounds targeting TRKs are currently being explored in clinical trials and, notably, one of these compounds, larotrectinib (VITRAKVI®), has received accelerated approval by the United States Food and Drug Administration (FDA) for adult and paediatric solid tumours with a NTRK fusion without known resistance mutations. In addition, entrectinib has received breakthrough designation status by the United States FDA for the treatment of cancers types harbouring NTRK fusions. Hence, there is an active interest in clinical oncology for NTRK fusions, which has prompted an urgent need to define the routine diagnostic test to identify gene fusions as a companion diagnostic method to support clinical decision in this context. Irrespective of the method adopted for NTRK detection, high activity of anti-NTRK agents and therefore the necessity to guarantee these agents to all NTRK+ patients, strongly supports a NTRK screening program for patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of any solid cancer
* Availability of tumor tissue for biomarker analyses (at least 5 slides, 4 micron)
* Signed informed consent form

Exclusion Criteria:

* No tumor tissue available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients with solid tumors, irrespective of tumor stage.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-02-05 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
To assess the incidence of NTRK rearrangements in patients with solid tumors in Italy | 36 months
  Tumor tissue slides (4 micron) will be tested for NTRK positivity by means of immunohistochemistry (IHC) and then confirmed by means of fluorescence in-situ hybridization (FISH).

SECONDARY OUTCOMES:
To define incidence of NTRK in different tumor types | 36 months
  The incidence of NTRK gene fusions across different tumor types involves determining how frequently these genetic alterations occur within various malignancies. This process is essential for understanding the potential role of targeted therapies, such as TRK inhibitors, in specific cancers

CONTACTS AND LOCATIONS:
Overall Officials: Federico Cappuzzo, PI, Principal Investigator — Fondazione FORT
Locations (2):
- Italy (2):
  - Grisel Maver Militello, Roma, RM
  - Istituti Fisioterapici Ospitalieri- Ifo - Istituto Regina Elena, Roma, RM